CLINICAL TRIAL: NCT06126718
Title: Phase I Randomized, Open-label, Parallel-controlled, Pharmacokinetic and Safety Study of BR201 Injection Versus Cosentyx in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR201-101
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BR201 (Experimental)
  Interventions: Drug: BR201
- Cosentyx (Secukinumab) (Active Comparator)
  Interventions: Drug: Cosentyx（Secukinumab ）

INTERVENTIONS:
Drug: BR201 — One-dosage on D1 and review pharmacokinetic and safety until D112 after drug given
  Arms: BR201
Drug: Cosentyx（Secukinumab ） — One-dosage on D1 and review pharmacokinetic and safety until D112 after drug given
  Arms: Cosentyx (Secukinumab)

SUMMARY:
This is a randomized, open-label, controlled Phase I study of BR201 administered by subcutaneous injection. This study will characterize the pharmacokinetic, safety and immunogenicity of BR201 versus Cosentyx（Secukinumab ） in healthy male subjects after a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent form；
* Healthy men 18-50 years of age at time of consent；
* Body weight of ≥50 kg and ≤ 80 kg and BMI ≥19 and ≤ 26 kg/m2.

Exclusion Criteria:

* Clinical laboratory examination results are abnormal and with clinical significance, or other clinical findings indicate diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, tumor, pulmonary, immune, mental or cardiovascular and cerebrovascular diseases) with clinical significance;
* Use of IL-17 or other monoclonal antibodies in the last 6 months;
* Positive for anti-IL-17 antibodies at screening;
* Evidence of tuberculosis infection;
* With active infection at screening or have been hospitalized for a serious infection during the 8 months prior to screening or use of antibiotics within 2 weeks of enrollment;
* Anti-IL-17 antibody active ingredient, excipients or latex allergy;
* With severe bleeding factors that affect venous blood collection or unwilling to undergo venipuncture;
* Use drug treatment (including prescription drugs, over-the-counter drugs, health product etc.) within 14 days before screening;
* Surgery within 2 months prior to screening; or plan to have surgery during the study period;.
* Have received live vaccines within 6 months prior to screening, or have used any vaccines within 4 weeks prior to screening, or plan to be vaccinated during the trial.;
* History of malignant neoplasms；
* Hepatitis B and/or Hepatitis C; or HIV antigen/antibody positive; or Treponema pallidum antibody positive; .
* Blood donation or massive blood loss (> 400 ml) within 3 months or blood loss (> 200 ml) within 1 month before signing the informed consent; or plan to donate blood during the trial;
* Have a history of drug or substance abuse before screening; or positive drug abuse test results on the day of check-in;
* Acute disease occurred or with concomitant medication from the screening to use of the study drug.;
* Have pregnancy plan or sperm donation plan during the whole trial period and within 6 months after the completion of the study;
* Other conditions considered inappropriate to be included in this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Till Day112
  Area under the cure from 0 to infinite
Cmax | Till Day112
  The max concentration after drug given

SECONDARY OUTCOMES:
AUC0-t | Till Day112
  Area under the cure from 0 to some time
Tmax | Till Day112
  The time for drug enlarge to max concentration
T1/2 | Till Day112
  Half life
Vz/F | Till Day112
  Apparent volume of distribution
CL/F | Till Day112
  Clearance
Immunogenicity | Till Day112
  ADA
AE | Till Day112
  Advance event
Evaluation about injection site reactions | 0 mins, 0.5 hours, 24 hours and 72 hours after drug given
  Evaluation about injection site reactions
ECG | Till Day112
  ECG
Incidence of laboratory abnormalities | Till Day112
  To be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China